CLINICAL TRIAL: NCT04926402
Title: Effectiveness of Kangaroo Care Education Programme on Mothers, Nurses, and Infants Outcomes in Neonatal Intensive Care Unit
Brief Title: Kangaroo Care Education Programme (KCEP)
Acronym: KCEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Sharmiza Samsudin, Principle Investigator, University of Malaya
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 201765-5310
Record Dates: First submitted 2021-05-19; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Kangaroo-Mother Care Method
Keywords: Kangaroo Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): The control group received standard routine care
- Kangaroo care education program (Experimental): The experimental group received a maternal kangaroo care education program
  Interventions: Other: Kangaroo Care Education Program

INTERVENTIONS:
Other: Kangaroo Care Education Program — It is a special method of caring for a premature infant in which the baby is positioned for at least 1 hour a day in an upright skin-to-skin and chest-to-chest contact with its mother.
  Arms: Kangaroo care education program

SUMMARY:
A quasi-experimental and longitudinal study was conducted to evaluate the effectiveness of the kangaroo care education program (KCEP) on Mothers, Nurses, and Infants Outcomes in a Neonatal Intensive Care Unit. Forty-eight mother-infant dyads were enrolled per arm in the control and experimental groups. The control group received standard routine care, while the experimental group received a maternal kangaroo care education program.

DETAILED DESCRIPTION:
Introduction:

Kangaroo care (KC) is a simple, low cost and highly effective evidence-based nursing intervention that can benefit from mother-infant bonding attachment. Most mothers of premature infants will experience stress being separated from their premature infants. Bonding with premature infants will develop their brain and also make them feel loved, safe, and secure. Therefore, KC will help in bonding attachment, increase weight gain, decrease hospitalization, and increase breastfeeding rates.

Aim:

This study aims to investigate the effectiveness of two programs; a nursing education program and a mother education program regarding KC techniques on mothers, nurses, and infant outcomes.

Method:

A combination of two designs: Quasi-experimental and longitudinal designs with self-administered questionnaires were carried out to evaluate mothers, nurses, and infant outcomes using the Kangaroo Care Questionnaires Survey (KCQs) and Parental Stressor Scale: Neonatal Intensive Care Unit, Parental and Relationship (PSS: NICU: P&R) at a neonatal intensive care unit (NICU) of a Malaysian teaching hospital in Klang Valley. The kangaroo care education program (KC-EP) included theoretical and practical sessions on the KC benefits and hands-on KC techniques. The study consisted of three phases: Phase I (n=48 mother-infants dyads) in the control group, Phase II (n=47 nurses - KC-EP), and Phase III (n=48 mother-infants dyads-KC-EP) in the experimental group. Data collection for mothers and infants occurred at various time points during the study; pre-intervention (T0) post - 1-month intervention (T1) and post - 3-month intervention (T2). For the nursing outcomes occurred before and after the 7th day of the intervention program. The results were analyzed using the Statistical Package of Social Sciences(SPSS) version 23. Descriptive statistics were used to analyze the demographic data and items of the questionnaire. GLM univariate and repeated measure analysis of variance (RM-ANOVA) followed by Bonferroni test for mean comparison between control and experimental groups at (T0, T1, and T2).

ELIGIBILITY:
Inclusion Criteria:

* Premature infant at corrected age between 28 weeks to 36+6 weeks gestation.
* Both mothers and premature infants were medically and surgically stable.
* Mothers were willing to perform KC and admitted to the NICU.

Exclusion Criteria:

* Surgical infant i.e cleft lip, cleft palate, spina bifida, exomphalos, and omphalocele.
* Infant required medical treatment eg. prolonged phototherapy treatment.
* Trisomy 21.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Mothers
Enrollment: 96 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline perceptions of KC at 1-month and 3-month among the mothers. | Baseline, 1-month, and 3- month.
  The respondents were asked to answer 20 items on perceptions of KC. A 5-point Likert scale was used (strongly disagree-1 to strongly agree-5). A lower mean score reflecting a better perception of KC.
Change from baseline knowledge of KC at 1-month and 3-month among the mothers. | Baseline, 1-month, and 3- month.
  The respondents were asked to answer 11 items on knowledge of KC. They were given 'true', 'false', and 'not sure' to indicate their knowledge of KC, with higher mean scores indicating a better level of knowledge
Change from baseline perceived barrier to KC at 1-month and 3-month among the mothers. | Baseline, 1-month, and 3- month.
  The respondents were asked to answer 19 items on perceived barriers to practicing KC. The scale ranged from very influential (5) to not influential at all (1). A lower mean score of perceived barriers means the mothers are very positive.
Change from baseline perceived stress at 1-month and 3-month among the mothers. | Baseline, 1-month, and 3- month.
  The respondents were asked to answer 19 items on perceived stress level. A 5-point Likert scale ranging from not at all stressful (1) to extremely stressful (5), to reflect the level of stress faced by mothers with their premature infant's admission into the NICU. The lower the mean stress scores reported by the mothers, the lower the stress level.
Change from baseline weight gain at 1-month and 3 month among infants. | Baseline, 1-month, and 3- month
  The infants' weight were measured and recorded.
Change in number of days of hospitalization among the infants. | From day of admission at 28 weeks of gestation until 44 weeks of hospitalization.
  The infants' days of hospitalization were recorded.
Change from baseline breast feeding status at 1-month and 3-month among the infants. | Baseline, 1-month and 3-month
  The breast feeding status of infants were recorded.
Change from baseline perceptions of KC at 1-month and 3-month among the nurses. | Baseline, 1-month and 3-month
  The respondents were asked to answer 20 items on perceptions of KC. A 5-point Likert scale was used (strongly disagree-1 to strongly agree-5). A lower mean score reflecting a better perception of KC.
Change from baseline knowledge of KC at 1-month and 3-month among the nurses. | Baseline, 1-month and 3-month
  The respondents were asked to answer 11 items on knowledge of KC. They were given 'true', 'false', and 'not sure' to indicate their knowledge of KC, with higher mean scores indicating a better level of knowledge.
Change from baseline practice of KC at 1-month and 3-month among the nurses. | Baseline, 1-month and 3-month
  Respondents were asked to answer 11 items on practice of KC. A 5-point Likert scale. The descriptors were: very uncomfortable (1), somewhat uncomfortable (2), neither comfortable (3), somewhat comfortable (4) and very comfortable (5). A lower mean score indicated a high level of confidence and skills in initiating KC.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmiza Samsudin, PhD, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper L, Morrill A, Russell RB, Gooding JS, Miller L, Berns SD. Close to me: enhancing kangaroo care practice for NICU staff and parents. Adv Neonatal Care. 2014 Dec;14(6):410-23. doi: 10.1097/ANC.0000000000000144. PMID 25422927
- [Background] Conde-Agudelo A, Diaz-Rossello JL. Kangaroo mother care to reduce morbidity and mortality in low birthweight infants. Cochrane Database Syst Rev. 2016 Aug 23;2016(8):CD002771. doi: 10.1002/14651858.CD002771.pub4. PMID 27552521
- [Background] Cho ES, Kim SJ, Kwon MS, Cho H, Kim EH, Jun EM, Lee S. The Effects of Kangaroo Care in the Neonatal Intensive Care Unit on the Physiological Functions of Preterm Infants, Maternal-Infant Attachment, and Maternal Stress. J Pediatr Nurs. 2016 Jul-Aug;31(4):430-8. doi: 10.1016/j.pedn.2016.02.007. Epub 2016 Mar 11. PMID 26975461
- [Result] Davanzo R, Brovedani P, Travan L, Kennedy J, Crocetta A, Sanesi C, Strajn T, De Cunto A. Intermittent kangaroo mother care: a NICU protocol. J Hum Lact. 2013 Aug;29(3):332-8. doi: 10.1177/0890334413489375. Epub 2013 Jun 4. PMID 23735714
- [Derived] Samsudin S, Chui PL, Ahmad Kamar A, Abdullah KL, Yu CW, Mohamed Z. The Impact of Structured Kangaroo Care Education on Premature Infants' Weight Gain, Breastfeeding and Length of Hospitalization in Malaysia. J Multidiscip Healthc. 2023 Apr 12;16:1023-1035. doi: 10.2147/JMDH.S403206. eCollection 2023. PMID 37077560

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT04926402/Prot_SAP_ICF_000.pdf